CLINICAL TRIAL: NCT01250470
Title: Phase I Study of Safety, Tolerability and Immunological Effects of SVN53-67/M57-KLH in Patients With Survivin-Positive Malignant Gliomas
Brief Title: Vaccine Therapy and Sargramostim in Treating Patients With Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 171010; NCI-2010-02042 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 171010 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2010-11-24; First posted 2010-11-30 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Oligoastrocytoma; Anaplastic Oligodendroglioma; Giant Cell Glioblastoma; Glioblastoma; Gliosarcoma; Mixed Glioma; Recurrent Brain Neoplasm
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (vaccine therapy) (Experimental): Patients receive Montanide ISA-51/survivin peptide vaccine SC followed by sargramostim SC on day 0. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  TREATMENT EXTENSION: After completion of study treatment, select patients may receive additional doses of Montanide ISA-51/survivin peptide vaccine SC and sargramostim SC. Treatment repeats every 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Montanide ISA-51/Survivin Peptide Vaccine; Biological: Sargramostim

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Montanide ISA-51/Survivin Peptide Vaccine — Given SC
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin

SUMMARY:
This phase I trial studies the side effects of vaccine therapy when given together with sargramostim in treating patients with malignant glioma. Vaccines made from survivin peptide may help the body build an effective immune response to kill tumor cells. Colony-stimulating factors, such as sargramostim, may increase the number of white blood cells and platelets found in bone marrow or peripheral blood. Giving vaccine therapy and sargramostim may be a better treatment for malignant glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicity profile of the SVN53-67/M57-KLH peptide in Montanide ISA 51 (Montanide ISA-51/survivin peptide vaccine) plus with GM-CSF (sargramostim).

SECONDARY OBJECTIVES:

I. To measure the immune responses induced by SVN53-67/M57-KLH with Montanide ISA 51 with GM-CSF.

TERTIARY OBJECTIVES:

I. To collect preliminary data on therapeutic efficacy of this combination against malignant glioma.

OUTLINE:

Patients receive Montanide ISA-51/survivin peptide vaccine subcutaneously (SC) followed by sargramostim SC on day 0. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at weeks 12, 16, 20, and 24.

TREATMENT EXTENSION: After completion of study treatment, select patients may receive additional doses of Montanide ISA-51/survivin peptide vaccine SC and sargramostim SC. Treatment repeats every 3 months in the absence of disease progression or unacceptable toxicity.

After completion of treatment extension, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of one of the following: glioblastoma multiforme, anaplastic astrocytoma, anaplastic oligodendroglioma or anaplastic mixed glioma or anaplastic oligoastrocytoma
* Must have recurrent or progressive disease following standard therapy
* Karnofsky performance status (KPS) greater than or equal to 70
* Human leukocyte antigen (HLA)-A *02 or HLA-A *03 blood cell haplotype documented by polymerase chain reaction (PCR) analysis or flow cytometry
* Survivin expression on patient's tumor cells documented by immunohistochemistry
* Must be free of systemic infection; subjects with active infections (whether or not they require antibiotic therapy) may be eligible after complete resolution of the infection; subjects on antibiotic therapy must be off antibiotics for at least 7 days before beginning treatment
* White blood count >= 3000/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 10.0 g/dL
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN)
* Total bilirubin =< 2.0 mg/dL
* Serum creatinine =< 1.5 x institutional upper limit of normal (ULN)
* Patients of child-bearing potential must agree to use acceptable contraceptive methods during treatment and for three months after its completion; women must have a negative serum pregnancy test
* Patients who have had recent cranial surgery are eligible for inclusion, but the vaccine may not be administered prior to post-operative day 14
* Patient or legal representative must be able to read, understand the investigational nature of this study and sign an Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Inability to obtain histologic proof of malignancy or material unavailable for survivin testing
* Systemic corticosteroid therapy > 12 mg of dexamethasone or equivalent per day at study entry; patient should be on stable dose
* HLA-A *02 or HLA-A *03 negative
* Active infection requiring treatment (including human immunodeficiency virus [HIV] infection)
* Any medical condition that, in the opinion of the principal investigator, would compromise the patient's ability to participate in the study; this includes chronic active hepatitis infection, immunodeficiency disease, concurrent neurological condition or autoimmune disease
* Any of the following: pregnant or nursing women, or women of childbearing potential or their sexual partners who are unwilling to employ effective contraception (condoms, diaphragm, birth control pills, injections, intrauterine device, surgical sterilization, subcutaneous implants or abstinence)
* Concurrent chemotherapy, immunotherapy, radiotherapy, radiosurgery, interferon (e.g. Intron-A), allergy desensitization injections; growth factors (e.g. Procrit, Aranesp, Neulasta), interleukins (e.g. Proleukin) or any investigational therapeutic medication
* Evidence of current drug or alcohol abuse or psychiatric impairment, which in the investigator's opinion will prevent completion of the protocol therapy or follow-up
* Use of any experimental drug for any reason within the 30 days, or standard of care drug therapy within 28 days prior to randomization, or failure to fully recover from hematological effects of prior chemotherapy
* Known allergy or hypersensitivity to keyhole limpet hemocyanin (KLH), GM-CSF or magnetic resonance imaging (MRI) contrast agent
* Life expectancy less than 4 months
* Any prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement; participants with mild arthritis requiring nonsteroidal anti-inflammatory drug (NSAID) medications will not be excluded
* Participants who have another cancer diagnosis will be ineligible, except for those with: squamous cell cancer of the skin without known metastasis, basal cell cancer of the skin without known metastasis, carcinoma in situ of the breast (ductal carcinoma in situ [DCIS] or lobular carcinoma in situ [LCIS]), carcinoma in situ of the cervix and any cancer without distant metastasis that has been treated successfully, without evidence of recurrence or metastasis for over 5 years
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the patient an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-09-05 (Actual); Primary Completion 2014-05-29 (Actual); Study Completion 2014-05-29 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity, assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4 | Up to 30 days post-treatment
  The maximum grade of toxicity for each category of interest will be recorded for each patient and the summary results will be tabulated by category and grade. In addition, descriptive statistics will be utilized to present the toxicity findings in the treatment extension group.

SECONDARY OUTCOMES:
Immune response, defined as a patient who has responded in either interferon gamma enzyme-linked immunosorbent spot (ELISPOT) or multimer assays | Up to 6 months post-treatment
  For both assays, time course and magnitude of responses will be plotted and data will be treated using mixed-effect modeling. In addition, Fisher's exact test will be used to determine whether ELISPOT and multimer responses are associated. Additional exploratory analyses will be done as appropriate, and will be data-driven; hypothesis testing is not anticipated. Results will be displayed in plots and tables. In addition, descriptive statistics will be utilized to present the immunological findings in the treatment extension group.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fenstermaker, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States